CLINICAL TRIAL: NCT01709903
Title: A 26-week Treatment Randomized, Double-blind, Double Dummy, Parallel-group Study to Assess the Efficacy and Safety of QVA149 (Indacaterol / Glycopyrronium Bromide) Compared to Fluticasone/Salmeterol in Patients With Moderate to Severe COPD
Brief Title: A 26-week Treatment Randomized, Double-blind, Double Dummy Study to Assess the Efficacy and Safety of QVA149
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A2331
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Fluticasone-Salmeterol Drug Combination; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QVA149 (Experimental): QVA149 110/50 µg o.d., delivered via a single-dose dry powder inhaler (SDDPI), consisting of a fixed dose combination of indacaterol 110µg and NVA237 50µg
  Interventions: Drug: QVA149; Drug: Placebo to fluticasone/salmeterol
- fluticasone/salmeterol (Active Comparator): Fluticasone/salmeterol 500/50 µg b.i.d., delivered via a dry powder inhaler Accuhaler® device
  Interventions: Drug: Fluticasone/salmeterol; Drug: Placebo to QVA149

INTERVENTIONS:
Drug: QVA149 — QVA149 110/50 µg capsules q.d. for inhalation, delivered via Novartis single dose dry powder inhaler (SDDPI).
  Other Names: Experimental: QVA149
  Arms: QVA149
Drug: Fluticasone/salmeterol — Active fluticasone/salmeterol (500/50µg) b.i.d via a dry power inhaler Accuhaler® device.
  Other Names: Comparator: Fluticasone/salmeterol
  Arms: fluticasone/salmeterol
Drug: Placebo to QVA149 — Placebo to QVA149 with SDDPI
  Other Names: Experimental: QVA149
  Arms: fluticasone/salmeterol
Drug: Placebo to fluticasone/salmeterol — Placebo to fluticasone/salmeterol with Accuhaler
  Other Names: Comparator: fluticasone/salmeterol
  Arms: QVA149

SUMMARY:
To demonstrate the non-inferiority of QVA149 110/50 µg o.d. to fluticasone/salmeterol 500/50 µg b.i.d. in terms of trough Forced Expiratory Volume in one second (FEV1) (mean of 23 hours 15 min and 23 hours 45 min post QVA149 dose) following 26 weeks of treatment in patients with moderate to severe COPD

DETAILED DESCRIPTION:
To demonstrate the non-inferiority of QVA149 110/50 µg o.d. to fluticasone/salmeterol 500/50 µg b.i.d. in terms of trough Forced Expiratory Volume in one second (FEV1) (mean of 23 hours 15 min and 23 hours 45 min post QVA149 dose) following 26 weeks of treatment in patients with moderate to severe COPD.

The study population will consist of approximate 736 male and female adults (age 40 years and greater) with a clinical diagnosis of stable COPD [GOLD (2010)] and a smoking history of at least 10 pack years. It is anticipated that approximately 981 patients will need to be screened in order to randomize 736 patients into 2 treatment arms of the study with an equal randomization ratio, meaning QVA149 (368 patients), fluticasone/salmeterol (368 patients). Treatment randomization will be stratified by current/ex-smoker status and prior ICS use. It is intended that 552 patients will complete the study at Week 26 without major protocol deviations. Dropouts will not be replaced.

This will be a multi-national study, including China, and at least two other countries.

Standardization FEV1 AUC0-12h will be performed in a subgroup of around 100 patients (50 patients per treatment arm) in pre-selected centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe stable COPD (Stage II or Stage III) according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guideline.

Current or ex-smokers who have a smoking history of at least 10 pack years. Patients with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) ≥ 30% and < 80% of the predicted normal, and post-bronchodilator FEV1/FVC < 0.7.

Modified Medical Research Council (mMRC) grade of at least 2 at Visit 2.

Exclusion Criteria:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive Human Chorionic Gonadotropin (hCG) laboratory test.

Patents with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia (BPH), bladder-neck obstruction, moderate to severe renal impairment or urinary retention. BPH patients who are stable on treatment can be considered.

Patients with a history of long QT syndrome or whose QTc measured at run-in (Visit 2) (Fridericia method) is prolonged (>450 ms for males and females) as confirmed by the central Electrocardiogram (ECG) assessor.

Patients with Type I or uncontrolled Type II diabetes. Patients who have not achieved spirometry result at Visit 2 in accordance with American Thoracic Society/European Respiratory Society (ATS/ERS) criteria for acceptability and repeatability.

Patients with, a) any history of asthma or, b) onset of respiratory symptoms prior to age 40 years.

Patients with concomitant pulmonary disease (e.g. lung fibrosis, primary bronchiectasis, sarcoidosis, interstitial lung disorder, pulmonary hypertension).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- Argentina (7):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Rojas, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Chile (2):
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
  - Novartis Investigative Site, Viña del Mar, Vina Del Mar
- China (20):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Jiangyin
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai
- Taiwan (6):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei County, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Lin-Ko

REFERENCES:
- [Derived] Zhong N, Wang C, Zhou X, Zhang N, Humphries M, Wang L, Patalano F, Banerji D. Efficacy and Safety of Indacaterol/Glycopyrronium (IND/GLY) Versus Salmeterol/Fluticasone in Chinese Patients with Moderate-to-Severe Chronic Obstructive Pulmonary Disease: The Chinese Cohort from the LANTERN Study. COPD. 2016 Dec;13(6):686-692. doi: 10.1080/15412555.2016.1182970. Epub 2016 Aug 11. PMID 27715335
- [Derived] Zhong N, Wang C, Zhou X, Zhang N, Humphries M, Wang L, Thach C, Patalano F, Banerji D; LANTERN Investigators. LANTERN: a randomized study of QVA149 versus salmeterol/fluticasone combination in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2015 Jun 5;10:1015-26. doi: 10.2147/COPD.S84436. eCollection 2015. PMID 26082625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized into 2 treatment arms of the study with an equal 1:1 randomization ratio: QVA149 and Flut/Salm
Pre-assignment Details: A total of 1189 patients were screened; 744 (62.6%) completed the screening phase while 445 (37.4%) patients discontinued prior to completion of the screening phase
Period: Overall Study
Arm/Group | QVA149 | Fluticasone/Salmeterol
Started | 372 (Randomized set) | 372 (Randomized set)
Completed | 343 | 333
Not Completed | 29 | 39
Not completed — administrative problems | 2 | 6
Not completed — Abnormal test procedure results | 1 | 0
Not completed — In ability to use device | 1 | 1
Not completed — no longer needed study drug | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 2 | 0
Not completed — Protocol Violation | 3 | 2
Not completed — Lack of Efficacy | 3 | 3
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Adverse Event | 11 | 18

BASELINE CHARACTERISTICS:
Population: Three patients in the Flut/Salm treatment arm: were excluded from the FAS, safety set and PPS as they were randomized in error and did not receive the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 | Fluticasone/Salmeterol | Total
Number analyzed (Participants) | 372 | 369 | 741
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Set
  years | 64.8 (7.82) | 65.3 (7.91) | 65.0 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Set
  Participants
    Female | 31 | 38 | 69
    Male | 341 | 331 | 672
Race (NIH/OMB) [Count of Participants; unit: Participants] — Safety Set
  Participants
    American Indian or Alaska Native | 1 | 2 | 3
    Asian | 314 | 309 | 623
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 55 | 58 | 113
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) Following 26 Weeks of Treatment to Demonstrate the Non-inferiority of QVA149 110/50 μg o.d. to Fluticasone/Salmeterol 500/50 μg b.i.d
Description: Measurement of QVA149 110/50 μg o.d. to fluticasone/salmeterol 500/50 μg b.i.d. in terms of trough FEV1 (mean of 23 h 15 min and 23 h 45 min post QVA149 dose) following 26 weeks of treatment in patients with moderate to severe COPD.
Time Frame: 26 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
liters | 1.248 (0.0173) | 1.176 (0.0172)

2. Secondary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) Following 26 Weeks of Treatment to Demonstrate the Superiority of QVA 110/50μg o.d. to Fluticasone/Salmeterol 500/50 μg b.i.d
Time Frame: 26 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
liters | 1.259 (.0170) | 1.183 (0.0168)

3. Secondary Outcome: Standardized Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 0-4 Hours
Description: Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) 0-4h at Day 1 was measured via spirometry conducted according to internationally accepted standards. Measurements were made at 0, 5, 15, and 30 minutes; and 1, 2, 3 and 4 hours post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. Mixed model used: AUC FEV1 = treatment + baseline FEV1 + FEV1 reversibility components + baseline smoking status + baseline ICS use + country + center (country) + error. Center was included as a random effect nested within country.
Time Frame: Day 1, 12 and 26 weeks
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
Liter
  Day 1 (n=369,364) | 1.317 (0.0096) | 1.252 (0.0094)
  12 weeks (n=350,338) | 1.388 (0.0163) | 1.262 (0.0161)
  26 weeks (n=339,323) | 1.351 (0.0167) | 1.229 (0.0167)

4. Secondary Outcome: Analysis of FEV1 (L) Trough Response (Pre-dose) Over the Whole Treatment Period
Description: Average of Trough Forced Expiratory Volume in one second (FEV1)
Time Frame: 6,12,18 and 26 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
liter
  Week 6 (n=356,341) | 1.256 (0.0151) | 1.184 (0.0149)
  week 12 (n=346,333) | 1.265 (0.0158) | 1.191 (0.0156)
  week 18 (n=339,332) | 1.252 (0.0166) | 1.174 (0.0164)
  week 26 (n=338,324) | 1.226 (0.0171) | 1.142 (0.0171)

5. Secondary Outcome: Analysis of Trough FVC (L) Over the Whole Treatment Period
Description: Average of Trough Forced Vital Capacity (FVC) at 23 hours 15 min and the 23 hours 45 min post dose
Time Frame: 12 and 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
liter
  Day 1 (n=350,351) | 3.040 (0.0288) | 2.957 (0.0280)
  Week 12 (n=342,332) | 3.036 (0.0304) | 2.835 (0.0302)
  week 26 (n= 333,323) | 2.966 (0.0334) | 2.793 (0.0333)

6. Secondary Outcome: Health Related Quality of Life Analysis of SGRQ Total Score After 26 Weeks of Treatment
Description: A Total and three component scores are calculated: Symptoms; Activity; Impacts. Each component of the questionnaire is scored separately:The score for each component is calculated separately by dividing the summed weights by the maximum possible weight for that component and expressing the result as a percentage: Score = 100 x Summed weights from all positive items in that component divided by Sum of weights for all items in that component The Total score is calculated in similar way: Score = 100 x Summed weights from all positive items in the questionnaire divided by Sum of weights for all items in the questionnaire Sum of maximum possible weights for each component and Total: Symptoms 566.2 Activity 982.9 Impacts 1652.8 Total (sum of maximum for all three components) 3201.9 The proportion of patients who achieve a clinically important improvement of at least 4 units in the total SGRQ will be analyzed. The higher the score the more symptoms of disease are present.
Time Frame: 26 weeks
Population: Full Analysis set
Measure: Mean (Standard Error); unit: numbers on a scale
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
numbers on a scale
  Week 26 (n= 340,329) | 31.20 (1.118) | 32.00 (1.118)
  Week 26 LOCF(n=354,342) | 31.74 (1.136) | 32.43 (1.130)

7. Secondary Outcome: Analysis of the TDI Focal Score Over the Whole Treatment Period
Description: The Transition Dyspnea Index (TDI) total score after 12 and 26 weeks of treatment will be analyzed using the same mixed model as specified for the primary analysis with the Baseline Dyspnea Index (BDI) total score as the baseline.Total score ranging - 9 to + 9. The lower the score, the more deterioration in severity of dyspnea. One additional option in each category, which does not contribute to the score, allows for circumstances in which impairment is due to reasons other than dyspnea. ."Baseline 12 weeks" and "Baseline 26 weeks", were the baseline scores for available participants analyzed for each time point.
Time Frame: 12 and 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Numbers on a scale
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
Numbers on a scale
  Baseline 12 weeks (n=348,337) | 6.36 (0.096) | 6.36 (0.104)
  12 weeks (n=348,337) | 2.62 (0.240) | 2.40 (0.238)
  Baseline 26 weeks (n=335,326) | 6.38 (0.097) | 6.40 (0.105)
  26 weeks (n=335,326) | 3.02 (0.266) | 2.86 (0.266)

8. Secondary Outcome: Rescue Medication Use: Summary of the Mean Daily, Daytime and Nighttime Number of Puffs of Rescue Medication, by 4 Weekly Intervals
Description: The number of puffs of rescue medication taken in the previous 12 hours will be recorded in the Patient Diary in the morning and evening. "Baseline 12 weeks" and "Baseline 26 weeks", were the baseline scores for available participants analyzed for each time point. Less puffs taken is better.
Time Frame: 12 and 26 weeks
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: # of puffs
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
# of puffs
  Baseline Daytime 12-16 weeks (n=329,318) | 1.57 (1.934) | 1.69 (2.130)
  Daytime 12-16 weeks (n=329,318) | 0.66 (1.185) | 0.61 (1.117)
  Baseline Nighttime 12-16 weeks (n=322,307) | 1.25 (1.5954) | 1.24 (1.707)
  Nighttime 12-16 weeks (n=322,307) | 0.52 (1.007) | 0.49 (0.960)
  Baseline Daytime 24-26 weeks (n=326,315) | 1.54 (1.885) | 1.70 (2.160)
  Daytime 24-26 weeks (n=326,315) | 0.63 (1.226) | 0.62 (1.135)
  Baseline Night time 24-26 weeks (n=320,304) | 1.23 (1.588) | 1.21 (1.702)
  Night time 24-26 weeks (n=320,304) | 0.52 (1.087) | 0.48 (0.923)

9. Secondary Outcome: Symptoms Reported Using E-diary Over 12 and 26 Weeks of Treatment
Description: Percentage of nights with 'no nighttime awakenings', percentage of days with 'no daytime symptoms', and percentage of 'days able to perform usual daily activities' over 26 weeks (FAS)
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: % days in study
Arm/Group | QVA149 | Fluticasone/Salmeterol
Number analyzed (Participants) | 372 | 369
% days in study
  % nights 'no nighttime awakenings' (n=336,322) | 67.57 (2.138) | 67.86 (2.101)
  % days with 'no daytime symptoms' (n=341,334) | 7.31 (1.466) | 10.22 (1.425)
  % days able perform daily activities (n=341,334) | 44.02 (2.200) | 42.16 (2.140)

ADVERSE EVENTS:
Groups:
- QVA149 110mcg/50mcg: QVA149 110/50 µg o.d., delivered via a single-dose dry powder inhaler (SDDPI), consisting of a fixed dose combination of indacaterol 110µg and NVA237 50µg
- Salmeterol/Fluticasone 50mcg/500mcg: Fluticasone/salmeterol 500/50 µg b.i.d., delivered via a dry powder inhaler Accuhaler® device
Arm/Group | QVA149 110mcg/50mcg | Salmeterol/Fluticasone 50mcg/500mcg
Serious Adverse Events (participants affected / at risk) | 20/372 | 35/369
Other Adverse Events (participants affected / at risk) | 107/372 | 135/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 110mcg/50mcg (N=372) | Salmeterol/Fluticasone 50mcg/500mcg (N=369)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 1 | 0
Cor pulmonale chronic (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Pterygium (Eye disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hyperplasia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 2 | 4
Septic shock (Infections and infestations) | 0 | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 110mcg/50mcg (N=372) | Salmeterol/Fluticasone 50mcg/500mcg (N=369)
Gastritis (Gastrointestinal disorders) | 0 | 4
Pyrexia (General disorders) | 3 | 5
Bronchitis (Infections and infestations) | 7 | 3
Nasopharyngitis (Infections and infestations) | 30 | 45
Pneumonia (Infections and infestations) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 13 | 26
Upper respiratory tract infection bacterial (Infections and infestations) | 5 | 3
Viral upper respiratory tract infection (Infections and infestations) | 1 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 69 | 83
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Hypertension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial